CLINICAL TRIAL: NCT03751293
Title: A Phase Ⅰ Study Evaluating Safety and Efficacy of C-CAR088 Treatment in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of BCMA-directed CAR-T Cells Treatment in Subjects With r/r Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0203-006
Record Dates: First submitted 2018-11-15; First posted 2018-11-23 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR088 (Experimental): Lymphocytes will be transduced with lentiviral vector containing CAR-BCMA gene
  Interventions: Biological: C-CAR088

INTERVENTIONS:
Biological: C-CAR088 — Autologous BCMA-directed CAR-T cells, single infusion intravenously at a target dose of 1.0-9.0 x 10^6 anti-BCMA CAR+ T cells/kg
  Other Names: CBM.BCMA Chimeric Antigen Receptor T cell

SUMMARY:
This is a single-center, non-randomized study to evaluate the safety and efficacy of C-CAR088 in relapsed or refractory multiple myeloma patient.

DETAILED DESCRIPTION:
The study will include the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation, Lymphodepleting Chemotherapy), C-CAR088 infusion and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate in this study and signed informed consent.
2. Age 18-70 years old, male or female.
3. Meet the internationally accepted Criteria for the diagnosis of multiple myeloma (IMWG diagnostic criteria 2014).
4. Patients with relapsed or refractory multiple myeloma who meet at least one of the following conditions:

   * Subjects must have received at least two therapy regimens (including proteasome inhibitor or immune-modulator therapy, disease progress or relapse after the last therapy).
   * Subjects have received only one therapy regimen, but the investigators judge that patients have unmet treatment needs or can't get benefit from current treatment options.
5. Subjects have one or more measurable multiple myeloma lesion, must include one of the following conditions:

   * Serum M protein≥1 g/dl(10g/L)
   * Urine M protein≥200 mg/24h
   * Serum free light chain(sFLC): κ/λ ratio abnormal and ≥10 mg/dl
6. Bone marrow sample is confirmed as BCMA-positive by flow cytometry or pathological examination.
7. At least 2 weeks from monoclonal antibody therapy prior to CAR T cell therapy.
8. ECOG scores 0 - 1.
9. Normal cardiac diastolic function, left ventricular ejection fraction (LVEF) ≥ 50% (detected by echocardiography), no serious arrhythmia.
10. No active pulmonary infections, normal pulmonary function and oxygen saturation ≥ 92% on room air.
11. No contraindications of leukapheresis.
12. Expected survival > 12 weeks.
13. Female subjects in childbearing age, their serum or urine pregnancy test must be negative,until 7 days before cell therapy and all subjects must agree to take effective contraceptive measures during the trial.

Exclusion Criteria:

1. Have a history of allergy to cellular products.
2. Any kind of these laboratory testing: including but not limited to,serum total bilirubin≧1.5mg/dl, serum ALT, AST≧2.5×ULN, serum creatinine≧2.0mg/dl, Hb (hemoglobin)<80g/L, neutrophils<1000/mm^3, platelets≦50000/mm^3 or platelet count maintained by transfusion.
3. Subjects with the following clinically significant cardiovascular diseases.
4. A history of craniocerebral trauma, consciousness disorder, epilepsy, severe cerebral ischemia or hemorrhagic disease.
5. Use any anticoagulant (except aspirin).
6. Patients requiring urgent treatment due to tumor progression or spinal cord compression.
7. Patients with CNS metastasis or symptoms of CNS involvement.
8. The investigators judge that any increase in the risk of the subject or interference with the results of the trial.
9. After allogeneic hematopoietic stem cell transplantation.
10. Plasma cell leukemia.
11. One week before leukapheresis and one week before CART cell infusion, treated with more than 5mg/d prednisone (or equal amount of other corticosteroids).
12. Subjects with any autoimmune disease or any immune deficiency disease or other disease in need of immunosuppressive therapy.
13. Uncontrolled active infection.
14. Prior treatment with CAR T therapy or any other genetically modified T cell therapy.
15. Live vaccine inoculation within four weeks before enrollment.
16. Hepatitis B or hepatitis C virus infection (including carriers), syphilis, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV-infected persons.
17. Have a history of alcoholism, drug addiction and mental illness.
18. Participated in any other clinical trial within three months.
19. The investigators believe that there are other circumstances that are not suitable for the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety: The incidence of treatment-emergent adverse events (TEAEs) | 30 days
  The incidence of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 months
Progression free survival (PFS) | 6 months, 12 months
The CART cell duration in vivo | 12 months
  The copys of BCMA-CART DNA in peripheral blood with qPCR method
The soluble BCMA changes in peripheral blood | 12 months
  The amount of soluble BCMA in peripheral blood with ELISA method

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China

REFERENCES:
- [Derived] Qu X, An G, Sui W, Wang T, Zhang X, Yang J, Zhang Y, Zhang L, Zhu D, Huang J, Zhu S, Yao X, Li J, Zheng C, Zhu K, Wei Y, Lv X, Lan L, Yao Y, Zhou D, Lu P, Qiu L, Li J. Phase 1 study of C-CAR088, a novel humanized anti-BCMA CAR T-cell therapy in relapsed/refractory multiple myeloma. J Immunother Cancer. 2022 Sep;10(9):e005145. doi: 10.1136/jitc-2022-005145. PMID 36100310